CLINICAL TRIAL: NCT06628310
Title: A Phase 2 Randomized Study to Evaluate the Safety, Efficacy, and Optimal Dose of Telisotuzumab Adizutecan in Combination With Fluorouracil, Leucovorin, and Budigalimab as First-Line Treatment in Subjects With Locally Advanced Unresectable or Metastatic Gastric, Gastroesophageal Junction, or Esophageal Adenocarcinoma (AndroMETa-GEA-977)
Brief Title: A Study to Evaluate the Adverse Events, Efficacy, and Optimal Dose of Intravenous (IV) ABBV-400 in Combination With IV Fluorouracil, Leucovorin, and Budigalimab in Adult Participants With Locally Advanced Unresectable or Metastatic Gastric, Gastroesophageal Junction, or Esophageal Adenocarcinoma
Acronym: AndroMETa-GEA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M24-977; 2024-513008-32 (Other: EU CT)
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Unresectable or Metastatic Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: Locally Advanced Unresectable or Metastatic Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma; ABBV-400; ABBV-181; Budigalimab; Telisotuzumab Adizutecan
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — budigalimab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Stage 1: Dose Escalation ABBV-400 (Experimental): Participants will receive escalating doses of telisotuzumab adizutecan (ABBV-400) in combination with a fixed dose of fluorouracil, leucovorin and budigalimab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Budigalimab; Drug: Fluorouracil; Drug: Leucovorin
- Stage 2 Arm 1: Dose Optimization ABBV-400 Dose A (Experimental): Participants will receive telisotuzumab adizutecan (ABBV-400) dose A in combination with a fixed dose of fluorouracil, leucovorin and budigalimab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Budigalimab; Drug: Fluorouracil; Drug: Leucovorin
- Stage 2 Arm 2: Dose Optimization ABBV-400 Dose B (Experimental): Participants will receive telisotuzumab adizutecan (ABBV-400) dose B in combination with a fixed dose of fluorouracil, leucovorin and budigalimab as part of the approximately 6 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Budigalimab; Drug: Fluorouracil; Drug: Leucovorin
- Stage 2 Arm 3: Dose Optimization Standard of Care (SOC) (Experimental): Participants will receive a fixed dose of leucovorin (folinic acid), fluorouracil, oxaliplatin (FOLFOX) and budigalimab as part of the approximately 6 year study duration.
  Interventions: Drug: Budigalimab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion
  Other Names: ABBV-400
  Arms: Stage 1: Dose Escalation ABBV-400; Stage 2 Arm 1: Dose Optimization ABBV-400 Dose A; Stage 2 Arm 2: Dose Optimization ABBV-400 Dose B
Drug: Budigalimab — IV Infusion
  Other Names: ABBV-181
Drug: Fluorouracil — IV Infusion; IV Injection
Drug: Leucovorin — IV Infusion; IV Injection
  Other Names: Folinic Acid
Drug: Oxaliplatin — IV Infusion
  Arms: Stage 2 Arm 3: Dose Optimization Standard of Care (SOC)

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess adverse events and change in disease activity when telisotuzumab adizutecan (ABBV-400) is given in combination with Fluorouracil, Leucovorin, and a programmed cell death receptor 1 (PD1) inhibitor Budigalimab. The combination (AFLB) will be given to adult participants to treat locally advanced unresectable or metastatic gastric, gastroesophageal junction, or esophageal adenocarcinoma (mGEA).

Telisotuzumab Adizutecan (ABBV-400) and Budigalimab are investigational drugs being developed for the treatment of mGEA. Fluorouracil and Leucovorin are drugs approved for the treatment of mGEA. This study will be divided into two stages, with the first stage treating participants with increasing doses of ABBV-400 within the AFLB regimen until the dose reached is tolerable and expected to be efficacious. Participants will then be randomized into groups called treatment arms where one group will receive Budigalimab and FOLFOX (Fluorouracil, Leucovorin, and Oxaliplatin) . A further two treatment groups will receive AFLB, but with two optimized doses of ABBV-400 to allow for the best dose to be studied in the future. Approximately 180 adult participants with mGEA will be enrolled in the study in 51 sites worldwide.

In the dose escalation stage, participants will be treated with increasing intravenous (IV) doses of telisotuzumab adizutecan (ABBV-400) within the AFLB regimen until the dose reached is tolerable and expected to be efficacious. In the dose optimization stage, participants will receive FOLFOX or receive AFLB, but with one of two optimized doses of ABBV-400. The study will run for a duration of approximately 6 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Have inoperable, advanced or metastatic histologically- or cytologically confirmed gastric, gastroesophageal junction, or esophageal adenocarcinoma.
* Have measurable disease determined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Human epidermal growth factor receptor 2 (HER2) negative disease, defined as immunohistochemistry (IHC) (0, or 1+) or fluorescence in situ hybridization (FISH) negative.
* Known programmed death ligand 1 (PD-L1) status at screening, or availability of tumor tissue for central PD-L1 testing prior to enrollment.

Exclusion Criteria:

* Have prior systemic therapy in the locally advanced, unresectable, or metastatic setting.
* History of clinically significant, intercurrent lung-specific illnesses including, but not limited to those listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by Investigator | Through Study Completion, Approximately 6 Years
  PFS is defined as the time from the first dose of study drug to the first occurrence of radiographic progression based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as determined by investigator or death from any cause, whichever occurs earlier.
Percentage of Participants with Objective Response (OR) as Assessed by Investigator | Through Study Completion, Approximately 6 Years
  OR is defined as confirmed complete response (CR) or confirmed partial response (PR) as assessed by investigator per RECIST version 1.1.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Disease Control (DC) as Assessed by Investigator | Through Study Completion, Approximately 6 Years
  DC is defined as best overall response of confirmed CR or confirmed PR, or stable disease (SD) (with a minimum duration of 14 weeks) based on RECIST, version 1.1 as determined by the investigator.
Duration of Response (DOR) as Assessed by Investigator | Through Study Completion, Approximately 6 Years
  DOR is defined as the time from the first documented CR or PR to the first occurrence of radiographic progression per RECIST version 1.1 as determined by investigator or death from any cause, whichever occurs first.
Overall Survival (OS) | Through Study Completion, Approximately 6 Years
  OS is defined as the time from first dose of study drug to the event of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (47):
- United States (7):
  - City of Hope National Medical Center /ID# 268690, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 272630, Irvine, California
  - UCLA - Santa Monica /ID# 270024, Santa Monica, California
  - AdventHealth Orlando /ID# 268561, Orlando, Florida
  - Hattiesburg Clinic /ID# 268572, Hattiesburg, Mississippi
  - Duke University Medical Center /ID# 268186, Durham, North Carolina
  - Millennium Research & Clinical Development /ID# 268540, Houston, Texas
- Belgium (3):
  - Algemeen Ziekenhuis klina /ID# 268754, Brasschaat, Antwerpen
  - Universitair Ziekenhuis Leuven /ID# 269957, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 270223, Liège
- Canada (3):
  - Princess Margaret Cancer Centre /ID# 268277, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM) /ID# 268763, Montreal, Quebec
  - Jewish General Hospital /ID# 268413, Montreal, Quebec
- China (5):
  - Beijing Cancer Hospital /ID# 268455, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences(Langfang) /ID# 277479, Langfang, Hebei
  - Harbin Medical University Cancer Hospital /ID# 268452, Harbin, Heilongjiang
  - Union Hospital - Tongji Medical College /ID# 268796, Wuhan, Hubei
  - The first Affiliated Hospital, Zhejiang University School of Medicine. /ID# 268782, Hangzhou, Zhejiang
- Germany (5):
  - Universitaetsklinikum Freiburg /ID# 270407, Freiburg im Breisgau, Baden-Wurttemberg
  - TUM Klinikum rechts der Isar /ID# 267792, Munich, Bavaria
  - Krankenhaus Nordwest /ID# 268462, Frankfurt am Main, Hesse
  - Universitaetsklinikum Leipzig /ID# 270432, Leipzig, Saxony
  - Haematologisch-Onkologische Praxis Eppendorf /ID# 268024, Hamburg
- Israel (5):
  - Meir Medical Center /ID# 267998, Kfar Saba, Central District
  - Soroka Medical Center /ID# 268301, Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 267755, Tel Aviv, Tel Aviv
  - Shaare Zedek Medical Center /ID# 267752, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 267753, Jerusalem
- Japan (5):
  - Aichi Cancer Center /ID# 268124, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 268083, Kashiwa-shi, Chiba
  - Shizuoka Cancer Center /ID# 268123, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 268648, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 268656, Koto-ku, Tokyo
- Pan American Center for Oncology Trials /ID# 268833, Rio Piedras, Puerto Rico
- Spain (4):
  - Hospital Universitario de Navarra /ID# 270119, Pamplona, Navarre
  - Hospital General Universitario Gregorio Maranon /ID# 270037, Madrid
  - Complexo Hospitalario Universitario de Ourense /ID# 270042, Ourense
  - Hospital Clínico Universitario de Valencia /ID# 270040, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 267672, Kaohsiung City
  - China Medical University Hospital /ID# 267667, Taichung
  - National Cheng Kung University Hospital /ID# 267669, Tainan
  - National Taiwan University Hospital /ID# 267666, Taipei
  - Taipei Veterans General Hospital /ID# 267664, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 267668, Taoyuan
- United Kingdom (3):
  - Barts Health NHS Trust /ID# 270796, London, Greater London
  - Oxford University Hospital NHS Trust /ID# 274614, Oxford, Oxfordshire
  - NHS Tayside Health Board /ID# 270799, Dundee

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-977